CLINICAL TRIAL: NCT03203928
Title: Effectiveness of a Tailored Occupational Therapy Intervention for Women With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Effectiveness of a Tailored Occupational Therapy Intervention for Women With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor of rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR4416
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Occupational Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Therapy for Women with ADHD (Experimental): 7-week tailored intervention for women with ADHD who have difficulty carrying out student, worker, spousal, and parenting roles due to poor time management, organization of their physical environments, management of internal and external stressors, and regulation of internal and external stimulation. Implementation of organizational, time management, stress management, and sensory regulation strategies for the home, school/work, and community environments.
  Interventions: Behavioral: Occupational Therapy Intervention for Women with ADHD
- Control (No Intervention): No treatment provided.

INTERVENTIONS:
Behavioral: Occupational Therapy Intervention for Women with ADHD — The intervention will run for 7 weeks and consist of the following 1-hour sessions. Each intervention session will be facilitated by two CUMC occupational therapy students in each participant's home environment (or another environment of the participant's choosing such as the work or school environment).
  Implementation of organizational, time management, stress management, and sensory regulation strategies for the home, school/work, and community environments.
  Arms: Occupational Therapy for Women with ADHD

SUMMARY:
Although woman are diagnosed with Attention-deficit hyperactivity disorder (ADHD) at a 1:3 ratio with men, recent research suggests that woman may experience the same levels of adult ADHD as men but are underdiagnosed because symptoms may be less severe and/or mistaken for anxiety and depression. Women with ADHD typically experience problems in managing worker, student, spousal, and parenting roles dues to disorganization, poor time management, difficulty regulating internal and external stressors, and difficulty maintaining daily schedules and routines. Intervention effectiveness research has largely focused on pharmacological treatment of ADHD symptoms; however, while such pharmacological treatment tends to enhance concentration and reduce motor restlessness, it does not address the skills needed to successfully carry out daily life roles and activities dependent upon time management, prioritization of tasks, and regulation of emotional responses within the home, school/work, and community environments. In this study, the investigators aim to determine whether a 7-week tailored occupational therapy intervention addressing organization, time management, stress management, and sensory regulation in the home, school/work, and community environments can increase satisfaction in desired daily life activities, and reduce ADHD symptoms and stress levels in women with ADHD.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is believed to be neurologically based and characterized by enduring attentional problems, motor restlessness, and cognitive and motor impulsivity that impact one's ability to function optimally in daily life activities. ADHD is commonly diagnosed in childhood at a prevalence rate of 11% and a male to female ratio of 3:1. The prevalence of adult ADHD varies from 4 to 6% and it is estimated that two-thirds of adult ADHD disorders are extensions of childhood ADHD. Researchers have suggested that the male to female prevalence ratio is inaccurate and that females experience ADHD at similar levels to males but are underdiagnosed. While boys with ADHD are often identified by their teachers because of motor impulsivity and inattention, girls with ADHD who may experience attentional problems and impulsivity without significant hyperactivity, may fail to be identified by teachers as needing evaluation and treatment. Some studies have found that female children and adolescents who experience the ADHD symptoms of inattention, disorganization, poor time management, and distractibility are more likely to be misdiagnosed with depression and anxiety. When depression and anxiety occur in children and adolescents with undiagnosed ADHD symptoms, they may result from the inability to manage ADHD symptoms as they impact functional performance in the home, school, and community.

Much of the research exploring ADHD has been devoted to children and adolescents. The research examining adult ADHD has thus far largely attempted to describe the phenomenon of adult ADHD. Research investigating intervention effectiveness for adult ADHD has primarily focused on pharmacological treatment. The small body of research examining non-pharmacological treatment has found moderate effectiveness for pharmacological intervention combined with cognitive behavioral therapy and psychoeducation.

Missing from this body of literature is research specifically examining interventions for women with ADHD, who present symptoms that are both overlapping with and unique from their male counterparts.

Studies have found that women with ADHD tend to have difficulty maintaining and succeeding in employment, school, and parenting and spousal roles. The ability to organize and implement tasks associated with each role, follow daily schedules and routines needed to support desired roles, prioritize and manage tasks in a timely manner, and regulate internal and external stressors to maintain consistent emotional responses may be difficult for with women with ADHD.

In this study, the investigators aim to provide a 7-week tailored intervention for women with ADHD who have difficulty carrying out student, worker, spousal, and parenting roles due to poor time management, organization of their physical environments, management of internal and external stressors, and regulation of internal and external stimulation.

This intervention effectiveness study will use randomization and control. Twenty-four women who self-report diagnoses of ADHD will be recruited to participate and randomly assigned to either the intervention group (n=12) or control group (n=12). The intervention group will receive the 6-week intervention; the control group will not receive intervention (bit will receive an organization toolkit at study end).

ELIGIBILITY:
Inclusion Criteria:

* Females aged 21-55 years
* English-speaking
* Self-reported ADHD

Exclusion Criteria:

* Severe co-morbid condition such as an eating disorder, major depression, bipolar disorder, schizophrenia spectrum disorder, or substance use disorder

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Difference in Score on World Health Organization Adult ADHD Self-Report Scale between pre- and post-intervention | baseline and 8 weeks
  18-item, 5-point Likert scale that requires 5 minutes to complete

SECONDARY OUTCOMES:
Difference in Score on Perceived Stress Scale between pre- and post-intervention | baseline and 8 weeks
  10-item, 5-point, self-report Likert scale that requires 5 minutes to complete
Difference in Score on Canadian Occupational Performance Measure | baseline and 8 weeks
  5-item, 10-point rating scale designed to be completed conjointly by a therapist and participant and takes approximately 10 minutes to complete

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mentaldisorders (5th ed.). Arlington, VA: American Psychiatric Publishing.
- [Background] Centers for Disease Control and Prevention. (2017). Attention-deficit/hyperactivity disorder (ADHD). Retrieved from https://www.cdc.gov/ncbddd/adhd/data.html
- [Background] Vande Voort JL, He JP, Jameson ND, Merikangas KR. Impact of the DSM-5 attention-deficit/hyperactivity disorder age-of-onset criterion in the US adolescent population. J Am Acad Child Adolesc Psychiatry. 2014 Jul;53(7):736-44. doi: 10.1016/j.jaac.2014.03.005. Epub 2014 Apr 23. PMID 24954823
- [Background] Jaconis M, Boyd SJ, Hartung CM, McCrea SM, Lefler EK, Canu WH. Sex differences in claimed and behavioral self-handicapping and ADHD symptomatology in emerging adults. Atten Defic Hyperact Disord. 2016 Dec;8(4):205-214. doi: 10.1007/s12402-016-0200-y. Epub 2016 Jun 21. PMID 27329539
- [Background] Coles EK, Slavec J, Bernstein M, Baroni E. Exploring the gender gap in referrals for children with ADHD and other disruptive behavior disorders. J Atten Disord. 2012 Feb;16(2):101-8. doi: 10.1177/1087054710381481. Epub 2010 Sep 13. PMID 20837979
- [Background] Quinn PO, Madhoo M. A review of attention-deficit/hyperactivity disorder in women and girls: uncovering this hidden diagnosis. Prim Care Companion CNS Disord. 2014;16(3):PCC.13r01596. doi: 10.4088/PCC.13r01596. Epub 2014 Oct 13. PMID 25317366
- [Background] Fredriksen M, Dahl AA, Martinsen EW, Klungsoyr O, Faraone SV, Peleikis DE. Childhood and persistent ADHD symptoms associated with educational failure and long-term occupational disability in adult ADHD. Atten Defic Hyperact Disord. 2014 Jun;6(2):87-99. doi: 10.1007/s12402-014-0126-1. Epub 2014 Feb 5. PMID 24497125
- [Background] Biederman J, Fried R, Tarko L, Surman C, Spencer T, Pope A, Grossman R, McDermott K, Woodworth KY, Faraone SV. Memantine in the Treatment of Executive Function Deficits in Adults With ADHD. J Atten Disord. 2017 Feb;21(4):343-352. doi: 10.1177/1087054714538656. Epub 2016 Jul 28. PMID 24970718
- [Background] Philipsen A, Jans T, Graf E, Matthies S, Borel P, Colla M, Gentschow L, Langner D, Jacob C, Gross-Lesch S, Sobanski E, Alm B, Schumacher-Stien M, Roesler M, Retz W, Retz-Junginger P, Kis B, Abdel-Hamid M, Heinrich V, Huss M, Kornmann C, Burger A, Perlov E, Ihorst G, Schlander M, Berger M, Tebartz van Elst L; Comparison of Methylphenidate and Psychotherapy in Adult ADHD Study (COMPAS) Consortium. Effects of Group Psychotherapy, Individual Counseling, Methylphenidate, and Placebo in the Treatment of Adult Attention-Deficit/Hyperactivity Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1199-210. doi: 10.1001/jamapsychiatry.2015.2146. PMID 26536057
- [Background] Fuller-Thomson E, Lewis DA, Agbeyaka SK. Attention-deficit/hyperactivity disorder casts a long shadow: findings from a population-based study of adult women with self-reported ADHD. Child Care Health Dev. 2016 Nov;42(6):918-927. doi: 10.1111/cch.12380. Epub 2016 Jul 20. PMID 27439337